CLINICAL TRIAL: NCT06102681
Title: Examination of the Effect of Early Mobilization on Postoperative Recovery, Pain, Quality of Life and Complication Development in Elective Minimally Invasive Spine Surgery
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: because of less patient
Sponsor: Duzce University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AtiyeErbas
Record Dates: First submitted 2023-10-21; First posted 2023-10-26 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2023-10

CONDITIONS: Spine Fusion; Lumbar Disc Herniation; Cervical Disc Disease
Keywords: quality of life; pain; minimal invasive surgery; ambulation; ERAS; recovery
MeSH Terms: conditions — Intervertebral Disc Displacement; Pain

STUDY DESIGN:
Intervention Model Description: all participants will assigned to two grup. one grup will be intervention the other will be control.
Who Masked: Participant
Masking Description: single
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): Patients who are in the control group will receive standard clinical care and these patient will be stand up 1. day after operation.
- experimental group (Experimental): Patients who are in the experimental group will receive standard clinical care and they will stand up 8. hours after operation.
  Interventions: Other: intervention group

INTERVENTIONS:
Other: intervention group — we will measure, consider and compare patients pain level, quality of life and recovery process. For these aims we will use numeric pain scale, nottingham health profile and postoperative recovery index.
  Arms: experimental group

SUMMARY:
Accelerated Postoperative Recovery (ERAS) is a multidisciplinary approach aimed at facilitating faster and more effective recovery for patients undergoing surgical procedures. The ERAS protocol encompasses specific measures implemented during the preoperative, intraoperative, and postoperative phases. Its goal is to enable patients to achieve better outcomes by reducing postoperative pain, complications, and hospital stays. The multimodal and multidisciplinary approach to patient care during the perioperative period includes a combination of evidence-based interventions designed to reduce the stress of surgery to maintain anabolic homeostasis and promote recovery.

This approach involves preparing patients for surgery through assessment and education, optimizing intraoperative management (such as minimally invasive surgery, pain control, and optimal fluid management), and expediting postoperative recovery (e.g., through early feeding and mobilization). Early mobilization is considered a crucial element of this approach and is strongly recommended as part of ERAS guidelines across various surgical disciplines.

Prolonged bed rest following surgical treatment has been associated with adverse outcomes, such as thromboembolism, pneumonia, muscle weakness, and loss of physical conditioning. If a patient does not have physical limitations in the postoperative period, early ambulation benefits in the preservation of respiratory, circulatory, musculoskeletal, and gastrointestinal system functions, as well as in reducing complications related to anesthesia and surgery. Ultimately, it accelerates recovery, enables early discharge, reduces hospital costs, and lightens the workload of healthcare professionals.

DETAILED DESCRIPTION:
Postoperative Accelerated Recovery (ERAS) is a multidisciplinary approach aimed at facilitating the faster and more effective recovery of patients undergoing surgical operations. The ERAS protocol encompasses specific measures implemented during the preoperative, intraoperative, and postoperative periods. Its objective is to ensure better outcomes for patients by reducing postoperative pain, complications, and the duration of hospital stays. The multimodal and multidisciplinary approach to patient care during the perioperative period includes a combination of evidence-based interventions aimed at reducing the stress of surgery to maintain anabolic homeostasis and promote recovery.

This includes preparing the patient for surgery through assessment and education, ensuring the best possible management during surgery (such as minimally invasive surgery, pain control, and optimal fluid management), and expediting postoperative recovery (for example, through early feeding and mobilization). Early mobilization is considered one of the most crucial elements of this approach and is strongly recommended as part of ERAS guidelines in many surgical disciplines.

Prolonged post-surgical bed rest has been associated with adverse outcomes such as thromboembolism, pneumonia, reduced muscle strength, and physical conditioning loss. If a patient does not have physical limitations in the postoperative period, early mobilization is beneficial in preserving respiratory, circulatory, musculoskeletal, and gastrointestinal system functions and in reducing complications related to anesthesia and surgery. Ultimately, it accelerates recovery, enables early discharge, and reduces hospital costs and the workload of healthcare professionals.

Despite the well-recognized importance of early mobilization in surgical procedures, it has been reported that compliance with mobilization goals is low, and those unable to achieve early postoperative mobilization are at a higher risk of complications. Reviewing the literature, it is observed that patients undergoing spinal surgery tend to avoid movement during the postoperative period due to experiencing intense pain before the surgery.

In this context, the aim of this study is to examine the impact of postoperative mobilization timing on patients' recovery status, pain levels, quality of life, and the development of complications following spinal surgery. The results obtained from the study are intended to be reported, thus contributing to the literature in this field and serving as a resource for future studies in this area.

ELIGIBILITY:
Inclusion Criteria:

* Elective minimal invasive spinal surgery patients

Exclusion Criteria:

* patients who is under 18 and over 65
* patients who have intubation tupe
* patients have mental disorders
* patients who underwent emergency surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2023-11-27 (Actual); Primary Completion 2024-05-06 (Actual); Study Completion 2024-09-15 (Estimated)

PRIMARY OUTCOMES:
Pain level | before operation and after 10 days operation
  we will use to measure patient pain level Numeric Pain Scale (NPS) several times. The intensity of pain will measure the area in which the individual mark between 0 (no pain) and 10 (worst pain i felt in my life).

SECONDARY OUTCOMES:
Life Quality | before operation and after 10 days operation
  we will use to measure quality of life of patients with Nottingham Health Profile. Thanks to survey we will compare to both group quality of life level. the survey is consist of six sub-dimention and thirty-eight item. the survey will use two times, first one will measure after first ambulation and the second one will measure after 10 days later.
recovery process | before operation and after 10 days operation
  we will use to measure post operative recovery index to me for patients recovery process. the questionnaire is consist of 5 sub-dimention and 25 item. the survey will use two times, first one will measure after first ambulation and the second one will measure after 10 days later.

CONTACTS AND LOCATIONS:
Locations (1):
- Duzce University Faculty of Health Science, Düzce, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided